CLINICAL TRIAL: NCT02096133
Title: Regulation of the Stress-axis by Vitamin D3 in Subjects With Multiple Sclerosis; a Double-blinded, Randomized, Placebo-controlled Study
Brief Title: Vitamin D3 and the Stress-axis in MS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: difficulties with inclusion
Sponsor: Academic MS Center Limburg (Other)
Responsible Party: Principal Investigator, Raymond Hupperts, Prof. R.M.M. Hupperts, MD, PhD, neurologist, Academic MS Center Limburg
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: EMR200109_635; 2014-000728-97 (EudraCT Number)
Record Dates: First submitted 2014-03-21; First posted 2014-03-26 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis, vitamin D, HPA-axis, cortisol
MeSH Terms: conditions — Multiple Sclerosis | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cholecalciferol (Experimental): Patients receive 1dd 100ug vitamin D3 (drops) for 16 weeks
  Interventions: Drug: Cholecalciferol
- Placebo comparator (Placebo Comparator): placebo drops during 16 weeks
  Interventions: Other: Placebo comparator

INTERVENTIONS:
Drug: Cholecalciferol — Vitamin D3 solution
  Other Names: Vigantol Oil
  Arms: Cholecalciferol
Other: Placebo comparator — Placebo comparator
  Arms: Placebo comparator

SUMMARY:
Patients with multiple sclerosis (MS) have an increased risk of developing a major depression. The investigators observed a protective effect of high vitamin D levels on the risk of depression in MS. This might be driven by the effect of vitamin D on the stress-axis. Therefore, the main goal of the present study is to assess whether high dose vitamin D supplementation results in a suppression of the stress-axis, as measured by decreased levels of cortisol.

DETAILED DESCRIPTION:
The lifetime incidence of a major depression in Multiple Sclerosis (MS) is 50%. (Patten et al. Neurology 2003; 61(11):1524-7) Our group reported a negative correlation between vitamin D status and depression score of the Hospital Anxiety and Depression Scale (HADS) in a cross-sectional dataset of Dutch MS patients. (Knippenberg et al. Acta Neurol Scand 2011; 124(3):171-5) This suggests an interaction between vitamin D and biological mechanisms affecting susceptibility to depression. Currently, we have two main hypotheses: 1) Vitamin D regulates the hypothalamic stress axis in MS. Based on our findings that cortisol releasing hormone (CRH)-positive hypothalamic neurons in the brains of MS patients stained positive for the vitamin D receptor (VDR) and 1,25(OH)2D-24-hydroxylase (24-OHase). (smolders et al. J Neuropathol Exp Neurol 2013;72(2):91-105) 2) Vitamin D affects T cell cytokine profile and hereby the odds of developing depression. Also in non-MS depressed patients increased levels of pro-inflammatory cytokines are detected (Maes et al. Metab Brain Dis 2009; 24: 27-53). Vitamin D3 has shown to be a potent promotor of T cell regulation both in vitro and in vivo. (Smolders et al. J Neuroimmunol 2008;194:7-17 and Smolders et al. PLoS One 2010;5:e15235) The main goal of this study is to assess whether supplementation of high doses vitamin D3 results in a suppression of saliva cortisol day-curves in subjects with multiple sclerosis, and we will explore whether the pro-inflammatory cytokine profile of T lymphocytes is regulated.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Relapsing Remitting MS
* At start of study > 6 weeks in clinical remission of disease
* Age > 18 years.
* Premenopausal
* Treated with either no immune-modulating treatment, or the currently registered MS modulating treatments: Interferon beta 1a (Rebif®), Interferon Beta 1b (Betaferon® or Avonex®), Glatiramer Acetate (Copaxone®), dimethylfumarate (Tecfidera®), teriflunomide (Aubagio®)) or fingolimod (Gilenya®).

Exclusion Criteria:

* Any contraindication to vitamin D according to Summary of Product Characteristics: Hypercalcaemia, hypervitaminosis D, nephrolithiasis, diseases or conditions resulting in hypercalcaemia and/or hypercalciuria (incl. primary hyperparathyroidism), severe renal impairment .
* Use of dexamethasone or other systemic glucocorticosteroids <2 months prior to first study visit
* Supplementation of >=1000 IU/d (25µg) vitamin D2 or D3
* Medical history of disturbed vitamin D/ calcium metabolism other than low intake
* Present clinical (major)depression
* Present treatment with anti-depressants, benzodiazepines, or neuroleptics.
* Treatment with high-dose dexamethasone for MS exacerbation during study.
* Pregnancy or the intention to become pregnant during the study period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-10-13; Primary Completion 2016-11-07 (Actual); Study Completion 2016-11-07 (Actual)

PRIMARY OUTCOMES:
The area under the curve (AUC) of the cortisol day curve | At baseline and after 16 weeks of supplementation.
  This number is constructed by combining the saliva cortisol levels at awakening, 11:00, 15:00, 20:00, and 22:00 hours (5 time-points).

SECONDARY OUTCOMES:
The slope of the cortisol day-curve | At baseline and after 16 weeks of supplementation
  The slope of the day-curve is the slope of the decrease of saliva cortisol measured throughout the cortisol day curve
The cortisol awakening response | At baseline and after 16 weeks of supplementation
  The awakening response is described by the rise in saliva cortisol from awakening to 60 minutes after awakening with respectively measurements at awakening, 15 minutes, 30 minutes, 45 minutes and 60 minutes (5 time-points).
Clinical outcomes on depression | At baseline and after 16 weeks of supplementation
  The clinical outcomes on depression will be measured by the depression sub-score of HADS and the FSSS fatigue score.
Efficacy of supplementation | At baseline and after 16 weeks of supplementation. Side effects will also be checked at 8 weeks of supplementation.
  To measure efficacy 25(OH)D levels will be measured.
Side effects | At baseline, after 8 and after 16 weeks
  Side effects will be measured after 8 and 16 weeks of treatment. Serum levels of calcium, albumin and creatinine will be determined, as well as calcium and creatinine levels in urine.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Hupperts, MD, PhD, Principal Investigator — Academic MS Center Limburg, Orbis MC
Locations (2):
- Netherlands (2):
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - Academic MS Center Limburg, Orbis Medical Center, Sittard-Geleen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rolf L, Damoiseaux J, Huitinga I, Kimenai D, van den Ouweland J, Hupperts R, Smolders J. Stress-Axis Regulation by Vitamin D3 in Multiple Sclerosis. Front Neurol. 2018 Apr 26;9:263. doi: 10.3389/fneur.2018.00263. eCollection 2018. PMID 29755397